CLINICAL TRIAL: NCT04325022
Title: Prospective, Multi-center Study to Evaluate the Safety and Effectiveness of the OR3O™ Dual Mobility System in Primary and Revision Total Hip Arthroplasty (THA) Procedures
Brief Title: Safety and Effectiveness Study of OR3O™ Dual Mobility System in THA
Acronym: OR3O
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OR3O.2019.08
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2024-11

CONDITIONS: Advanced Degeneration of the Hip Joint; Revision of the Hip Joint
Keywords: OR3O; THA; Dual Mobility; hip revision; hip replacement; hip joint; hip implant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Primary Total Hip Arthroplasty (THA): OR3O Dual Mobility System used in primary THA
  Interventions: Device: Primary Total Hip Arthroplasty
- Revision Total Hip Arthroplasty (THA): OR3O Dual Mobility System used in revision THA
  Interventions: Device: Revision Total Hip Arthroplasty

INTERVENTIONS:
Device: Primary Total Hip Arthroplasty — Primary Total Hip Arthroplasty using the OR3O Dual Mobility System in combination with compatible components
  Groups: Primary Total Hip Arthroplasty (THA)
Device: Revision Total Hip Arthroplasty — Revision Total Hip Arthroplasty using the OR3O Dual Mobility System in combination with compatible components
  Groups: Revision Total Hip Arthroplasty (THA)

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the OR3O™ Dual Mobility System. The study will evaluate the outcome of the Total Hip Arthroplasty using the OR3O™ Dual Mobility System over a ten year period. Survivorship of THA will be assessed up to ten years.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Subject is a suitable candidate for implanting the OR3O™ Dual Mobility System in primary or revision total hip replacement in the Investigator's judgement.
* Subject is skeletally mature in the Investigator's judgement.
* Subject is 18 - 80 years old (inclusive).
* Subject has any of the following conditions:

  * Advanced degeneration of the hip joint as a result of degenerative, post-traumatic, or rheumatoid arthritis (RA);
  * Fracture or avascular necrosis of the femoral head;
  * Failure of previous hip surgery: joint reconstruction, internal fixation, arthrodesis, hemiarthroplasty, surface replacement arthroplasty, or total hip replacement;
  * All forms of osteoarthritis (OA);
  * Patients with hips at risk of dislocation;
  * Femoral neck fracture or proximal hip joint fracture.
* Subject provides written informed consent for study participation using an Independent Ethical Committee (IEC) / Institutional Review Board (IRB) approved consent form before any study procedures are performed, including pre-operative data review and/or collection of data on electronic Case Report Forms (eCRFs).
* Subject is willing and able to participate in required follow-up visits and is able to complete study activities.
* Subject has all required study pre-operative and operative data available in their medical record for collection if consent is given after their THA surgery.

Revision Subjects:

* Subject has a REDAPT™ Modular Shell implanted which does not require revision or will receive a REDAPT™ Modular Shell during revision THA.
* Subject has a S+N compatible stem which does not require revision or will receive a S+N compatible stem during revision THA.

Exclusion Criteria:

All subjects:

* Subject has conditions that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately-sized implant, e.g.:

  * blood supply limitations;
  * insufficient quantity or quality of bone support, e.g., osteoporosis, metabolic disorders which may impair bone formation, radioactive bone disease, tumor around hip joint, and osteomalacia;
  * infections or other conditions which may lead to increased bone resorption.
* Subject has dysplasia of hip joint with CROWE Grade III, IV.
* Subject has bodily disease(s) that may interfere with THA survival or outcome.
* Subject has life expectancy of less than 10 years.
* Subject has mental or neurological conditions which impair the subject's ability or willingness to restrict activities that may put the affected limb at risk.
* Subject has physical conditions or activities which tend to place extreme loads on implants, e.g., Charcot joints, muscle deficiencies, multiple joint disabilities.
* Subject has neuromuscular dysfunctions (paralysis, myolysis and abductor muscle weakness) which will cause unstable hip joint or abnormal gait after surgery.
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study.
* Subject has an active infection - systemic or at the site of intended surgery.
* Subject has a Body Mass Index > 40.0 kg/m².
* Subject has a known allergy to any component of the devices used in the study.
* Subject is pregnant or breast feeding.
* Subject is entered in another investigational drug, biologic, or device study within 30 days of active study participation.

Revision Subjects:

* Subject has inadequate implant support with an increased risk of implant failure if support is not achieved, poor bone quality exists, or smaller sized implants are utilized.
* Subject needs revision of a fractured ceramic head or liner.
* Subject was already enrolled into this study as primary THA case.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is a suitable candidate for implanting the OR3O™ Dual Mobility System in primary or revision total hip replacement in the Investigator's judgement
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Survivorship of Primary Total Hip Arthroplasty (THA) | 2 years
  Assess survivorship of the OR3O™ Dual Mobility System at 2 years post implantation in Primary THA procedures. Survivorship is defined as no revision of the Acetabular Implant and OR3O™ Liner.

SECONDARY OUTCOMES:
Survivorship of individual Total Hip Arthroplasty (THA) components (OR3O Dual Mobility, acetabular shell, femoral head) | up to 10 years
  Survivorship of the following specific components will be presented individually: OR3O™Dual Mobility System, Acetabular Shell, Femoral head. The endpoint of interest is time to occurrence of a revision of the specific component due to any reason.
Harris Hip Score (HHS) | Pre-Op, 6 weeks, 6 months, 1 year, 2 years, 5 years, and 10 years
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Total scores range from 0 (worst) to 100 (best). The total scores and scores for each of the domains will be presented. The modified Harris Hip Score (mHHS) includes all the same domains as the HHS except for the hip range of motion (2 items, 0-5 points). Total mHHHs scores range from 0 (worst) to 95 (best). The total mHHS score maybe used in place of the total HHS score.
Five-level EuroQol five-dimensional (EQ-5D-5L) score | Pre-Op, 6 weeks, 6 months, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale. The descriptive system is used to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas.
  The visual analogue scale records the subject's self-rated health on a vertical visual analogue scale.The endpoints on the scale are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.
Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR.) | Pre-Op, 6 weeks, 6 months, 1 year, 2 years, 3 years, 5 years, 7 years, and 10 years
  The HOOS JR. is a short-form survey based on the Hip Disability and Osteoarthritis Outcome Score (HOOS) that specifically focuses on the outcome after THA. HOOS JR. consists of 2 areas: pain (2 items) and function, daily living (4 items). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes - no, mild, moderate, severe, extreme) and each question gets a score from 0 to 4. An interval score from 0-100 (0 indicating total hip disability and 100 indicating perfect hip health) is calculated (15).
Forgotten Joint Score 12 (FJS-12) | Pre-Op, 6 weeks, 6 months, 1 year, 2 years, 5 years, and 10 years
  The Forgotten Joint Score 12 (FJS-12) is a self-administered score where subjects are asked to rate their awareness of their hip arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced hip joint during the activities of daily living (i.e., higher score is a better outcome).
Radiographic Assessment - Acetabular Cup Migration | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Acetabular Cup Migration will be assessed from radiographs with the following definitions:
  0 - Absent: No evidence of acetabular cup migration ≥ 3 mm from baseline
  1 - Present: Presence of acetabular cup migration ≥ 3mm from baseline
Radiographic Assessment - Femoral Stem Subsidence | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Femoral Stem Subsidence will be assessed from radiographs with the following definitions:
  0 - Absent: No evidence of inferior movement of the femoral stem ≥ 3mm.
  1 - Present: Presence of inferior movement of the femoral stem compared to previously available imaging ≥ 3mm.
Radiographic Assessment - Osseointegration Status - Acetabular Cup | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Osseointegration Status - Acetabular Cup will be assessed from radiographs with the following definitions:
  0 - Absent: Absence of all radiographic signs or presence of only one radiographic sign of acetabular cup osseointegration
  1. - Partial: Presence of two radiographic signs of acetabular cup osseointegration.
  2. - Complete: Presence of three or more radiographic signs of acetabular cup osseointegration.
Radiographic Assessment - Acetabular Cup Loosening | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Acetabular Cup Loosening will be assessed from radiographs with the following definitions:
  0 - Absent: No evidence of specific imaging features of loosening at the acetabular bone-implant interface including significant radiolucency or change in position of the acetabular cup indicating a loss of fixation.
  1 - Present: Presence of apparent imaging features of loosening at the acetabular bone-implant interface including significant radiolucency or change in position of the acetabular cup indicating a loss of fixation.
Radiographic Assessment - Device Integrity | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Device Integrity will be assessed from radiographs with the following definitions:
  0 - Intact: No evidence of fracture, breakage or disassembly of any device component.
  1 - Failed: Presence of fracture, breakage or disassembly of one or more device components.
Radiographic Assessment - Progressive Radiolucency Acetabular Zones | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Progressive Radiolucency in all acetabular zones will be assessed from radiographs with the following definitions:
  0 - None: No evidence of an increase in width of the radiolucency > 1 mm
  1 - Present: Presence of an increase in width of the radiolucency > 1 mm
Radiographic Assessment - Progressive Radiolucency Femoral Zones | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Progressive Radiolucency in all femoral zones will be assessed from radiographs with the following definitions:
  0 - None: No evidence of an increase in width of the radiolucency > 1 mm
  1 - Present: Presence of an increase in width of the radiolucency > 1 mm
Radiographic Assessment - Osteolysis - Acetabular Cup | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Osteolysis Acetabular Cup will be assessed from radiographs with the following definitions:
  0 - None: No evidence of a ballooning / scalloping, progressive, periacetabular, bony destructive lesion with a maximum dimension > 5mm.
  1 - Present: Presence of a ballooning / scalloping, progressive, periacetabular, bony destructive lesion with a maximum dimension > 5mm.
Radiographic Assessment - Osteolysis - Femoral Stem | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Osteolysis Femoral Stem will be assessed from radiographs with the following definitions:
  0 - None: No evidence of a ballooning / scalloping, progressive, perifemoral, bony destructive lesion with a maximum dimension > 5mm.
  1 - Present: Presence of a ballooning / scalloping, progressive, perifemoral, bony destructive lesion with a maximum dimension > 5mm.
Radiographic Assessment - Anatomic Fracture | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Anatomic Fracture will be assessed from radiographs with the following definitions:
  0 - Absent: No evidence of anatomic fracture or other related complication.
  1 - Present: One or more of the following conditions are present: pelvic bone fracture or femoral bone fracture.
Radiographic Assessment - Heterotopic Ossification | 6 weeks, 1 year, 2 years, 5 years, and 10 years
  Heterotopic Ossification will be assessed from radiographs with the following definitions:
  0 - None: No evidence of heterotopic bone formation
  1. - Grade 1: (Class I) Islands of bone within the soft tissue about the hip
  2. - Grade 2: (Class II) Bone spurs from the pelvis or proximal end of the femur, leaving at least a centimeter between opposing bone surfaces.
  3. - Grade 3: (Class III) Bone spurs from the pelvis or proximal end of the femur, reducing the space between opossing bone surfaces to less than 1 cm.
  4. - Grade 4: (Class IV) apparent bone ankylosis of the hip

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — NYU Langone Health
Locations (12):
- United States (6):
  - University of Kentucky, Lexington, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - St. David's Center for Hip and Knee Replacement, Austin, Texas
- Australia (3):
  - Mater Health Services, Brisbane, Queensland
  - Royal Perth Hospital, Perth, Western Australia
  - Calvary John James Hospital, Deakin
- Canada (2):
  - South Health Campus, Calgary, Calgary, Alberta
  - St Michael's Hospital, Toronto, Ontario
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes